CLINICAL TRIAL: NCT02097849
Title: An Open-Label Study to Assess the Immune Response to Vaccination in Tecfidera® (BG00012)-Treated Versus Interferon-Treated Subjects With Relapsing Forms of Multiple Sclerosis.
Brief Title: Vaccination Response in Tecfidera-Treated Versus Interferon-Treated Participants With Relapsing Forms of Multiple Sclerosis.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 109MS307
Record Dates: First submitted 2014-03-25; First posted 2014-03-27 (Estimated); Results first posted 2017-06-02 (Actual); Last update posted 2017-06-02 (Actual); Status verified 2017-04

CONDITIONS: Relapsing Forms of Multiple Sclerosis
Keywords: vaccine; pneumococcal; meningococcal; tetanus diphtheria; immune response
MeSH Terms: interventions — Dimethyl Fumarate; Diphtheria-Tetanus Vaccine; 23-valent pneumococcal capsular polysaccharide vaccine; Meningococcal Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Non-Pegylated IFN Treated Plus Vaccinations (Active Comparator): Participants on a stable approved dose of a non pegylated IFN for ≥3 months will receive 3 vaccinations on Day 1 intramuscularly in the specified order:
  Td 0.5 mL PPSV23 0.5 mL MCV4 0.5 mL
  Interventions: Biological: tetanus diphtheria toxoids vaccine; Biological: 23-valent pneumococcal polysaccharide vaccine; Biological: meningococcal polysaccharide diphtheria conjugate vaccine (quadrivalent); Drug: non-pegylated interferon
- Tecfidera Treated Plus Vaccinations (Experimental): Participants on a stable approved dose of Tecfidera (240 mg BID) for ≥6 months will receive 3 vaccinations on Day 1 intramuscularly in the specified order:
  Td 0.5 mL PPSV23 0.5 mL MCV4 0.5 mL
  Interventions: Drug: dimethyl fumarate; Biological: tetanus diphtheria toxoids vaccine; Biological: 23-valent pneumococcal polysaccharide vaccine; Biological: meningococcal polysaccharide diphtheria conjugate vaccine (quadrivalent)

INTERVENTIONS:
Drug: dimethyl fumarate — Throughout the study participants will remain on their existing, stable dosing regimen of Tecfidera.
  Other Names: DMF; BG00012; Tecfidera
  Arms: Tecfidera Treated Plus Vaccinations
Biological: tetanus diphtheria toxoids vaccine — Administered as described in the treatment arm
  Other Names: Td; Tenivac
Biological: 23-valent pneumococcal polysaccharide vaccine — Administered as described in the treatment arm
  Other Names: Pneumovax 23; PPSV23
Biological: meningococcal polysaccharide diphtheria conjugate vaccine (quadrivalent) — Administered as described in the treatment arm
  Other Names: MCV4; Menveo
Drug: non-pegylated interferon — Throughout the study participants will remain on their existing, stable dosing regimen of non-pegylated IFN.
  Other Names: IFN
  Arms: Non-Pegylated IFN Treated Plus Vaccinations

SUMMARY:
Primary objective is to evaluate the immune response to vaccination with tetanus diphtheria toxoids vaccine (Td) in participants with relapsing forms of Multiple Sclerosis (MS) who have been treated with Tecfidera (BG00012) versus those treated with non pegylated interferon (IFN).

Secondary objective is to evaluate the immune response to vaccination with 23-valent pneumococcal polysaccharide vaccine (PPSV23) [a mostly T cell-independent humoral response] and meningococcal polysaccharide diphtheria conjugate vaccine, quadrivalent (MCV4) [T cell-dependent neoantigen response].

ELIGIBILITY:
Key Inclusion Criteria:

* Must have a confirmed diagnosis of relapsing remitting MS per the 2010 McDonald criteria.
* Must have a known tetanus immunization history with most recent tetanus vaccination given 2 to 15 years prior to Screening and an anti-tetanus serum immunoglobulin titer at Screening that is less than or equal to one-half the upper limit of detection for the assay.
* Must have been on a stable approved dose of Tecfidera (240 mg twice daily [BID]) [Group 1] for ≥6 months or on a stable approved dose of a non-pegylated IFN (e.g., Avonex, Betaseron, Rebif, Extavia) [Group 2] for ≥3 months prior to Day 1.

Key Exclusion Criteria:

* Clinical relapse requiring treatment within 30 days prior to Day 1.
* Pneumococcal vaccination within 5 years prior to Screening.
* Previous exposure to meningococcal vaccines.
* Known hypersensitivity to Td, PPSV23, or MCV4 or their components.

NOTE: Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2015-02-28 (Actual); Primary Completion 2016-05-02 (Actual); Study Completion 2016-05-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (14):
- United States (14):
  - Research Site, Gilbert, Arizona
  - Research Site, Thornton, Colorado
  - Research Site, Fort Lauderdale, Florida
  - Research Site, Sarasota, Florida
  - Research Site, Indianapolis, Indiana
  - Research Site, Lexington, Kentucky
  - Research Site, Auburn, Maine
  - Research Site, New York, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Akron, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Round Rock, Texas
  - Research Site, San Antonio, Texas

REFERENCES:
- [Derived] von Hehn C, Howard J, Liu S, Meka V, Pultz J, Mehta D, Prada C, Ray S, Edwards MR, Sheikh SI. Immune response to vaccines is maintained in patients treated with dimethyl fumarate. Neurol Neuroimmunol Neuroinflamm. 2017 Nov 15;5(1):e409. doi: 10.1212/NXI.0000000000000409. eCollection 2018 Jan. PMID 29159204

RESULTS

PARTICIPANT FLOW:
Groups:
- Non-Pegylated IFN Treated Plus Vaccinations: Participants on a stable approved dose of a non pegylated IFN for ≥ 3 months received 3 vaccinations on Day 1 intramuscularly in the specified order: Td 0.5 mL; PPSV23 0.5 mL; MCV4 0.5 mL.
- Tecfidera Treated Plus Vaccinations: Participants on a stable approved dose of Tecfidera (240 mg BID) for ≥ 6 months received 3 vaccinations on Day 1 intramuscularly in the specified order: Td 0.5 mL; PPSV23 0.5 mL; MCV4 0.5 mL.
Period: Overall Study
Arm/Group | Non-Pegylated IFN Treated Plus Vaccinations | Tecfidera Treated Plus Vaccinations
Started | 33 | 38
Completed | 33 | 38
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Non-Pegylated IFN Treated Plus Vaccinations | Tecfidera Treated Plus Vaccinations | Total
Number analyzed (Participants) | 33 | 38 | 71
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.7 (7.77) | 45.9 (6.10) | 45.3 (6.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 34 | 61
  Male | 6 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Tetanus Responders (≥ 2-Fold Rise) at Day 28 Compared to Prevaccination Level
Description: Percentage of participants with a ≥ 2-fold rise in anti-tetanus serum immunoglobulin G (IgG) levels (responders) from prevaccination to 4 weeks after Td vaccination.
Time Frame: Up to Week 4 (Day 28) postvaccination
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Non-Pegylated IFN Treated Plus Vaccinations | Tecfidera Treated Plus Vaccinations
Number analyzed (Participants) | 33 | 38
percentage of participants | 73 [54 to 87] | 68 [51 to 82]
Statistical Analysis 1: Comparison: Non-Pegylated IFN Treated Plus Vaccinations vs Tecfidera Treated Plus Vaccinations; Test type: Superiority or Other; p = 0.692, Clopper-Pearson Exact; Difference in proportion = -0.04, 95% CI 2-sided [-0.27 to 0.19]

2. Secondary Outcome: Percentage of Tetanus Responders (≥ 4-Fold Rise) at Day 28 Compared to Prevaccination Level
Description: Percentage of participants with a ≥ 4-fold rise in anti-tetanus serum IgG levels (responders) from prevaccination to 4 weeks after Td vaccination.
Time Frame: Up to Week 4 (Day 28) postvaccination
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Non-Pegylated IFN Treated Plus Vaccinations | Tecfidera Treated Plus Vaccinations
Number analyzed (Participants) | 33 | 38
percentage of participants | 61 [42 to 77] | 42 [26 to 59]
Statistical Analysis 1: Comparison: Non-Pegylated IFN Treated Plus Vaccinations vs Tecfidera Treated Plus Vaccinations; Responders at Day 28; Test type: Superiority or Other; p = 0.120, Clopper-Pearson Exact; Difference in proportion = -0.19, 95% CI 2-sided [-0.41 to 0.05]

3. Secondary Outcome: Percentage of Pneumococcal Serotype 3 (≥ 2-Fold Rise) Responders Compared to Prevaccination Level
Description: Percentage of participants with a ≥ 2-fold rise in anti-pneumococcal serum IgG levels against serotype 3 from prevaccination to 4 weeks (28 days) after PPSV23 vaccination.
Time Frame: Up to Week 4 (Day 28) postvaccination
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Non-Pegylated IFN Treated Plus Vaccinations | Tecfidera Treated Plus Vaccinations
Number analyzed (Participants) | 33 | 38
percentage of participants | 79 [61 to 91] | 66 [49 to 80]
Statistical Analysis 1: Comparison: Non-Pegylated IFN Treated Plus Vaccinations vs Tecfidera Treated Plus Vaccinations; Test type: Superiority or Other; p = 0.225, Clopper-Pearson Exact; Difference in proportions = -0.13, 95% CI 2-sided [-0.35 to 0.10]

4. Secondary Outcome: Percentage of Pneumococcal Serotype 3 (≥ 4-Fold Rise) Responders Compared to Prevaccination Level
Description: Percentage of participants with a ≥ 4-fold rise in anti-pneumococcal serum IgG levels against serotype 3 from prevaccination to 4 weeks (28 days) after PPSV23 vaccination.
Time Frame: Up to Week 4 (Day 28) postvaccination
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Non-Pegylated IFN Treated Plus Vaccinations | Tecfidera Treated Plus Vaccinations
Number analyzed (Participants) | 33 | 38
percentage of participants | 70 [51 to 84] | 47 [31 to 64]
Statistical Analysis 1: Comparison: Non-Pegylated IFN Treated Plus Vaccinations vs Tecfidera Treated Plus Vaccinations; Test type: Superiority or Other; p = 0.057, Clopper-Pearson Exact; Difference in proportions = -0.22, 95% CI 2-sided [-0.44 to 0.01]

5. Secondary Outcome: Percentage of Pneumococcal Serotype 8 (≥ 2-Fold Rise) Responders Compared to Prevaccination Level
Description: Percentage of participants with a ≥ 2-fold rise in anti-pneumococcal serum IgG levels against serotype 8 from prevaccination to 4 weeks (28 days) after PPSV23 vaccination.
Time Frame: Up to Week 4 (Day 28) postvaccination
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Non-Pegylated IFN Treated Plus Vaccinations | Tecfidera Treated Plus Vaccinations
Number analyzed (Participants) | 33 | 38
percentage of participants | 88 [72 to 97] | 95 [82 to 99]
Statistical Analysis 1: Comparison: Non-Pegylated IFN Treated Plus Vaccinations vs Tecfidera Treated Plus Vaccinations; Test type: Superiority or Other; p = 0.300, Clopper-Pearson Exact; Difference in proportions = 0.07, 95% CI 2-sided [-0.16 to 0.30]

6. Secondary Outcome: Percentage of Pneumococcal Serotype 8 (≥ 4-Fold Rise) Responders Compared to Prevaccination Level
Description: Percentage of participants with a ≥ 4-fold rise in anti-pneumococcal serum IgG levels against serotype 8 from prevaccination to 4 weeks (28 days) after PPSV23 vaccination.
Time Frame: Up to Week 4 (Day 28) postvaccination
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Non-Pegylated IFN Treated Plus Vaccinations | Tecfidera Treated Plus Vaccinations
Number analyzed (Participants) | 33 | 38
percentage of participants | 85 [68 to 95] | 82 [66 to 92]
Statistical Analysis 1: Comparison: Non-Pegylated IFN Treated Plus Vaccinations vs Tecfidera Treated Plus Vaccinations; Test type: Superiority or Other; p = 0.714, Clopper-Pearson Exact; Difference in proportions = -0.03, 95% CI 2-sided [-0.26 to 0.20]

7. Secondary Outcome: Percentage of Meningococcal Serogroup C Responders (≥ 2-Fold Rise) Compared to Prevaccination Level
Description: Percentage of participants with a ≥ 2-fold rise in anti-meningococcal serum IgG levels against serotype C from prevaccination to 4 weeks after MCV4 vaccination.
Time Frame: Up to Week 4 (Day 28) postvaccination
Population: One participant in the IFN group did not have an assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Non-Pegylated IFN Treated Plus Vaccinations | Tecfidera Treated Plus Vaccinations
Number analyzed (Participants) | 32 | 38
percentage of participants | 53 [35 to 71] | 53 [36 to 69]
Statistical Analysis 1: Comparison: Non-Pegylated IFN Treated Plus Vaccinations vs Tecfidera Treated Plus Vaccinations; Test type: Superiority or Other; p = 0.967, Clopper-Pearson Exact; Difference in proportions = 0, 95% CI 2-sided [-0.24 to 0.23]

8. Secondary Outcome: Percentage of Meningococcal Serogroup C Responders (≥ 4-Fold Rise) Compared to Prevaccination Level
Description: Percentage of participants with a ≥ 4-fold rise in anti-meningococcal serum IgG levels against serotype C from prevaccination to 4 weeks after MCV4 vaccination.
Time Frame: Up to Week 4 (Day 28) postvaccination
Population: One participant in the IFN group did not have an assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Non-Pegylated IFN Treated Plus Vaccinations | Tecfidera Treated Plus Vaccinations
Number analyzed (Participants) | 32 | 38
percentage of participants | 38 [21 to 56] | 37 [22 to 54]
Statistical Analysis 1: Comparison: Non-Pegylated IFN Treated Plus Vaccinations vs Tecfidera Treated Plus Vaccinations; Test type: Superiority or Other; p = 0.955, Clopper-Pearson Exact; Difference in proportions = -0.01, 95% CI 2-sided [-0.24 to 0.22]

9. Secondary Outcome: Ratio of Serum Tetanus Level at Day 28 to Prevaccination
Description: Median serum titer ratios from prevaccination to 4 weeks after Td vaccination.
Time Frame: Up to Week 4 (Day 28) postvaccination
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Non-Pegylated IFN Treated Plus Vaccinations | Tecfidera Treated Plus Vaccinations
Number analyzed (Participants) | 33 | 38
ratio | 6.128 [2.828 to 8.139] | 4.463 [1.955 to 8.244]

10. Secondary Outcome: Ratio of Serum Pneumococcal Antibodies (Serotype 3) Level at Day 28 to Prevaccination
Description: Median serum titer ratios from prevaccination to 4 weeks after PPSV23 vaccination.
Time Frame: Up to Week 4 (Day 28) postvaccination
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Non-Pegylated IFN Treated Plus Vaccinations | Tecfidera Treated Plus Vaccinations
Number analyzed (Participants) | 33 | 38
ratio | 9.667 [4.537 to 18.000] | 4.741 [2.000 to 11.000]

11. Secondary Outcome: Ratio of Serum Pneumococcal Antibodies (Serotype 8) Level at Day 28 to Prevaccination
Description: Median serum titer ratios from prevaccination to 4 weeks after PPSV23 vaccination.
Time Frame: Up to Week 4 (Day 28) postvaccination
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Non-Pegylated IFN Treated Plus Vaccinations | Tecfidera Treated Plus Vaccinations
Number analyzed (Participants) | 33 | 38
ratio | 27.000 [12.750 to 49.286] | 13.845 [6.000 to 28.250]

12. Secondary Outcome: Ratio of Serum Meningococcal Antibodies (Serogroup C) Level at Day 28 to Prevaccination
Description: Median serum titer ratios from prevaccination to 4 weeks after MCV4 vaccination.
Time Frame: Up to Week 4 (Day 28) postvaccination
Population: One participant in the IFN group did not have an assessment.
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Non-Pegylated IFN Treated Plus Vaccinations | Tecfidera Treated Plus Vaccinations
Number analyzed (Participants) | 32 | 38
ratio | 3.300 [1.000 to 11.159] | 3.408 [1.000 to 8.600]

13. Secondary Outcome: Number of Participants Experiencing Vaccination-Emergent Adverse Events (AEs) and Serious AEs
Description: An AE was any untoward medical occurrence that did not necessarily have a causal relationship with this treatment. A serious AE was any untoward medical occurrence that at any dose: resulted in death; was life-threatening; required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity; resulted in a congenital anomaly/birth defect; any other medically important event that, in the opinion of the Investigator, could have jeopardized the participant or required intervention to prevent one of the other outcomes listed in the definition above.
Time Frame: Day 1 to Week 4
Population: Participants who received at least one vaccination.
Measure: Number; unit: participants
Arm/Group | Non-Pegylated IFN Treated Plus Vaccinations | Tecfidera Treated Plus Vaccinations
Number analyzed (Participants) | 33 | 38
participants
  Any Event | 18 | 16
  Moderate or Severe Event | 9 | 7
  Severe Event | 2 | 0
  Event Related to Existing Therapy | 3 | 3
  Serious Event | 0 | 0
  Serious Event Related to Existing Therapy | 0 | 0
  Serious Event Related to Td Vaccine | 0 | 0
  Serious Event Related to PPSV23 Vaccine | 0 | 0
  Serious Event Related to MCV4 Vaccine | 0 | 0
  Withdrew From Study Due to an Event | 0 | 0

14. Secondary Outcome: Number of Participants With Shifts From Baseline in Hematology
Description: Shift to low includes normal to low, high to low, and unknown to low. Shift to high includes normal to high, low to high, and unknown to high.
Time Frame: Screening to Week 4
Population: n=participants whose baseline value was not low (or high) and who had at least one postbaseline value.
Measure: Number; unit: participants
Arm/Group | Non-Pegylated IFN Treated Plus Vaccinations | Tecfidera Treated Plus Vaccinations
Number analyzed (Participants) | 33 | 38
participants
  Hemoglobin: Shift to Low; n=28, 36 | 1 | 0
  Hemoglobin: Shift to High; n=32, 38 | 0 | 0
  Hematocrit: Shift to Low; n=31, 37 | 2 | 1
  Hematocrit: Shift to High; n=32, 38 | 0 | 0
  Red Blood Cell Count: Shift to Low; n=25, 32 | 1 | 4
  Red Blood Cell Count: Shift to High; n=33, 37 | 0 | 0
  White Blood Cell Count: Shift to Low; n=27, 30 | 2 | 4
  White Blood Cell Count: Shift to High; n=33, 38 | 2 | 0
  Neutrophils: Shift to Low; n=27, 34 | 3 | 2
  Neutrophils: Shift to High; n=33, 37 | 2 | 0
  Basophils: Shift to Low; n=33, 38 | 0 | 0
  Basophils: Shift to High; n=33, 38 | 0 | 0
  Monocytes: Shift to Low; n=33, 38 | 0 | 2
  Monocytes: Shift to High; n=33, 38 | 2 | 0
  Lymphocytes: Shift to Low; n=33, 22 | 4 | 1
  Lymphocytes: Shift to High; n=33, 38 | 0 | 0
  Eosinophils: Shift to Low; n=33, 38 | 0 | 0
  Eosinophils: Shift to High; n=33, 38 | 0 | 0
  Platelet Count: Shift to Low; n=31, 38 | 1 | 0
  Platelet Count: Shift to High; n=32, 37 | 0 | 0

15. Secondary Outcome: Number of Participants With Shifts From Baseline in Blood Chemistry
Description: as for outcome 14
Time Frame: Screening to Week 4
Population: n=participants whose baseline value was not low (or high) and who had at least one postbaseline value.
Measure: Number; unit: participants
Arm/Group | Non-Pegylated IFN Treated Plus Vaccinations | Tecfidera Treated Plus Vaccinations
Number analyzed (Participants) | 33 | 38
participants
  Alanine Aminotransferase: Shift to Low; n=33, 38 | 0 | 0
  Alanine Aminotransferase: Shift to High; n=30, 35 | 2 | 1
  Aspartate Aminotransferase: Shift to Low; n=33, 37 | 0 | 0
  Aspartate Aminotransferase: Shift to High; n=33,36 | 1 | 0
  Total Bilirubin: Shift to Low; n=32, 37 | 0 | 1
  Total Bilirubin: Shift to High; n=33, 38 | 0 | 0
  Gamma-glutamyl Transferase: Shift to Low; n=33, 38 | 0 | 0
  Gamma-glutamyl Transferase: Shift to High; n=33,38 | 0 | 0
  Blood Urea Nitrogen: Shift to Low; n=33, 38 | 0 | 0
  Blood Urea Nitrogen: Shift to High; n=33, 38 | 1 | 1
  Creatinine: Shift to Low; n=33, 38 | 0 | 0
  Creatinine: Shift to High; n=33, 37 | 0 | 0
  Sodium: Shift to Low; n=33, 38 | 0 | 0
  Sodium: Shift to High; n=33, 38 | 0 | 0
  Potassium: Shift to Low; n=33, 38 | 0 | 0
  Potassium: Shift to High; n=33, 38 | 0 | 0
  Chloride: Shift to Low; n=33, 38 | 1 | 0
  Chloride: Shift to High; n=33, 38 | 0 | 0

16. Secondary Outcome: Number of Participants With Abnormalities in Vital Signs
Description: Temperature increase: > 38 celcius (C) or ≥ 1 C increase from baseline. Pulse increase: > 120 beats per minute (bpm) or > 20 bpm increase from baseline. Pulse decrease: < 50 bpm or > 20 bpm decrease from baseline. Systolic blood pressure (SBP) increase: > 180 millimeters of mercury (mmHg) or > 40 mmHg from baseline. SBP decrease: < 90 mmHg or > 30 mmHg decrease from baseline. Diastolic blood pressure (DBP) increase: > 105 mmHg or > 30 mmHg increase from baseline. DBP decrease: < 50 mmHg or > 20 mmHg decrease from baseline.
Time Frame: Screening to Week 4
Population: Participants who had a baseline assessment and at least one postbaseline assessment.
Measure: Number; unit: participants
Arm/Group | Non-Pegylated IFN Treated Plus Vaccinations | Tecfidera Treated Plus Vaccinations
Number analyzed (Participants) | 32 | 38
participants
  Temperature Increase | 0 | 0
  Pulse Increase | 1 | 1
  Pulse Decrease | 0 | 0
  SBP Increase | 1 | 0
  SBP Decrease | 0 | 0
  DBP Increase | 0 | 1
  DBP Decrease | 0 | 0

ADVERSE EVENTS:
Time Frame: SAEs: Screening (Within 28 Days Before Day 1) up to Week 4 (Day 28 ±3 Days) or Early Withdrawal. AEs: Day 1 up to Week 4 (Day 28 ±3 Days) or Early Withdrawal
Description: Vaccination-emergent adverse events are presented.
Arm/Group | Non-Pegylated IFN Treated Plus Vaccinations | Tecfidera Treated Plus Vaccinations
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/38
Other Adverse Events (participants affected / at risk) | 14/33 | 11/38
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Non-Pegylated IFN Treated Plus Vaccinations (N=33) | Tecfidera Treated Plus Vaccinations (N=38)
Injection site erythema (General disorders) | 4 | 5
Injection site pain (General disorders) | 7 | 8
Injection site swelling (General disorders) | 3 | 3
Injection site warmth (General disorders) | 0 | 2
Pain (General disorders) | 3 | 1
Pyrexia (General disorders) | 2 | 2
Urinary tract infection (Infections and infestations) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Headache (Nervous system disorders) | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.